CLINICAL TRIAL: NCT06621303
Title: Autonomous Regulatory Monocytes (OPM Cells) for the Treatment of Diabetic Foot in a Single-arm Open-label Clinical Study
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Collaborators: Faendrich (Shanghai) Biotechnology Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DFTXB-2024-003
Record Dates: First submitted 2024-09-29; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-Arm, Open-Label Clinical Study Protocol for the Treatment of Diabetic Foot with Autoregulator (Experimental)
  Interventions: Biological: Diabetic foot ulcer treatment

INTERVENTIONS:
Biological: Diabetic foot ulcer treatment — The trial is designed to last up to 26 weeks, including a screening period of 1 week, a treatment period of 1 week, and an observation period of 24 weeks. According to the inclusion criteria, 10 diabetic patients with ulcers will be clinically screened, and after signing the informed consent form, they will be assigned a number. Post-injection of OPM cells, wound assessments are conducted weekly, with physical examinations and vital signs (pulse, blood pressure) recorded at weeks 4, 8, 12, 16, 20, and 24. Clinical laboratory tests (routine blood tests, tumor markers, etc.) are performed at week 12. Vascular CTA and immune cell count in wound lavage fluid are conducted at week 24 post-cellular intervention, followed by a final examination at week 24.

SUMMARY:
To reduce the risk of critical limb ischemia (CLI) in diabetic patients, repair local ulcers in the limbs of diabetic patients, and avoid the occurrence of amputation, Academician Van der Rijt has developed autoregulatory monocytes (OPM cells). These are derived from monocytes extracted from the peripheral blood of the patient, cultured in vitro using cytokines, which endow them with the capability to promote angiogenesis and tissue repair. Preliminary animal experiments and European clinical studies have shown that injecting OPM cells into the muscle around diabetic ulcers increases the paracrine of proteins related to angiogenesis and tissue recovery, promotes the regeneration and repair of tissue structure and function, and activates precursor cells or naive cells (including tissue-oriented stem cells) that are dormant or suppressed within tissues and organs. These cells replace and reconstruct the cells and tissues that have been damaged and lost function due to disease, thereby restoring physiological functions.

To explore whether this therapy can repair local ulcers in the limbs of diabetic patients, Shanghai Oriental Hospital, in collaboration with Van der Rijt (Shanghai) Biotechnology Co., Ltd., has initiated this exploratory clinical study to evaluate the safety and preliminary efficacy of OPM cells in the treatment of diabetic ulcers.

Study Objective： As a clinical study initiated by researchers, this study aims to explore the safety and preliminary efficacy of OPM cells in reducing complications in diabetic foot patients. The study will evaluate the potential of OPM cells to improve critical limb ischemia (CLI) and promote wound healing in diabetic foot ulcers.

Study Overall Design： The trial is designed to last up to 26 weeks, including a screening period of 1 week, a treatment period of 1 week, and an observation period of 24 weeks.

According to the inclusion criteria, 10 diabetic patients with ulcers will be clinically screened, and after signing the informed consent form, they will be assigned a number. Before treatment, measurements will be taken of the size of the ulcer wound, the immune cell count of the ulcer exudate, and vascular CTA detection, among others, and recorded.

On day 0, a clean and tidy single room will be arranged as the treatment room. Venous blood will be drawn from each participant sequentially, 200ml per participant, and then cultured in the cell laboratory for 4 days according to their assigned numbers. On day 4, samples will be taken for endotoxin, bacterial and mycoplasma testing, cell counting, and flow cytometry analysis. Once approved, OPM cells will be collected and suspended in 5% human serum albumin. The harvested OPM cells will be stored at 2~8°C and transported to the hospital. Upon arrival at Shanghai Oriental Hospital, sample testing will be conducted first. Only after the samples pass testing will the patients receive intramuscular injections. The OPM cells must be injected into the muscle around the ulcer within 6 hours after leaving the laboratory.

Wound assessments will be conducted weekly after injection. Physical examinations and vital signs (pulse, blood pressure) will be recorded at weeks 4, 8, 12, 16, 20, and 24. Clinical tests (blood routine, tumor markers, etc.) will be performed at week 12. Vascular CTA and immune cell count in wound lavage fluid will be detected at week 24 after cell intervention, and a final examination will be conducted at week 24.

The safety and efficacy of OPM cells in treating diabetic ulcer patients will be determined based on the healing of the wound size, the increase in the number of immune cells in the wound lavage fluid, and the increase in vascular collateral circulation.

ELIGIBILITY:
Inclusion Criteria:

* (1) Meet the diagnostic criteria for diabetes; (2) Present with clinical symptoms of lower limb ischemia; (3) Ancillary tests suggest lower extremity vascular disease. ABI <0.9 at rest, or ABI >0.9 at rest but symptoms of lower limb discomfort occur during exercise, with a decrease in ABI of 15%-20% after a treadmill test or imaging indicates vascular stenosis. If ABI cannot be measured, TBI can be used as a supplementary test, with TBI <0.7 indicating lower extremity vascular disease.

  (4) Male or female adult patients 18 years of age or older (including 18 years). Women of childbearing potential are allowed to be enrolled on the condition that:
* The pregnancy test is negative at the screening visit
* They agree to use appropriate contraceptive measures routinely before and during the study
* They agree not to attempt to become pregnant and not to breastfeed during the study. Women without childbearing potential are defined as postmenopausal for at least one year or surgically sterilized.

  (5) Diabetic patients with ulcers, where the ulcer surface area is between 2cm×2cm and 4cm×4cm.

  (6) Diabetic foot with Wagner grade II or below, including grade II. (7) Patients with ulcers that have not healed for more than one month. (8) Patients who voluntarily accept cell therapy. (9) After the nature of the study and data disclosure have been explained to the patient, the patient voluntarily signs a written informed consent form and agrees to participate in the study.

Patients with diabetic foot ulcers selected based on the inclusion criteria are classified as having mild ulcers.

Exclusion Criteria:

* (1) Ulcer surface area is less than 2cm×2cm or larger than 4cm×4cm; (2) Diabetic foot with Wagner grade higher than 3, including grade 3; (3) Ulcer onset within 1 month; (4) Patients requiring amputation; (5) Patients with diabetic foot complicated by severe infection; (6) Patients who are HIV positive, syphilis positive, or have active hepatitis B or C virus; (7) Patients with a history of alcohol abuse and/or drug use; (8) Pregnant or lactating mother patients; (9) Patients with malignant tumors or a history of malignant tumors; (10) Patients who are simultaneously participating in or planning to participate in any other clinical studies; (11) Patients with psychiatric or emotional issues; (12) Patients unwilling or unable to provide informed consent; (13) Patients with their own blood system diseases; (14) Patients who have previously had a diabetic foot amputation and have developed a new ulcer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of serious adverse reactions | During the 24 week follow-up period after treatment

SECONDARY OUTCOMES:
Ulcer wound size score | During the 24 week follow-up period after treatment
Score for the number of collateral vessels | During the 24 week follow-up period after treatment
Immune cell count score | During the 24 week follow-up period after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Berndt R, Hummitzsch L, Hess K, Albrecht M, Zitta K, Rusch R, Sarras B, Bayer A, Cremer J, Faendrich F, Gross J. Allogeneic transplantation of programmable cells of monocytic origin (PCMO) improves angiogenesis and tissue recovery in critical limb ischemia (CLI): a translational approach. Stem Cell Res Ther. 2018 Apr 27;9(1):117. doi: 10.1186/s13287-018-0871-8. PMID 29703251
- [Background] Broichhausen C, Riquelme P, Ahrens N, Wege AK, Koehl GE, Schlitt HJ, Banas B, Fandrich F, Geissler EK, Hutchinson JA. In question: the scientific value of preclinical safety pharmacology and toxicology studies with cell-based therapies. Mol Ther Methods Clin Dev. 2014 Jul 16;1:14026. doi: 10.1038/mtm.2014.26. eCollection 2014. PMID 26015968